CLINICAL TRIAL: NCT03116256
Title: The Effect of Very Low Calorie Diet (VLCD) With and Without Concomitant Resistance Exercise Training (RET) or High Intensity Interval Training (HIIT) on Muscle Protein Synthesis (MPS) in Middle-aged Overweight Male.
Brief Title: The Effect of Very Low Calorie Diet With and Without Exercise on Muscle Synthesis in Middle-aged Overweight Male.
Acronym: VLCDex
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Nottingham (Other)
Collaborators: University of Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: B12092016
Record Dates: First submitted 2017-03-31; First posted 2017-04-17 (Actual); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — High-Intensity Interval Training; Resistance Training

STUDY DESIGN:
Intervention Model Description: Participant will be randomised into one of the following group:
  1. VLCD (N=12),
  2. VLCD + RET (N=12)
  3. VLCD + HIIT (N=12)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- VLCD only (Other): Very low calorie diet (VLCD) only group- participants in this group will receive complete meal replacement for 6 weeks.
  Interventions: Dietary Supplement: Very low calorie diet (VLCD)
- VLCD+RET (Active Comparator): VLCD+RET group- participants in this group will receive complete meal replacement for 6 weeks and resistance exercise training 3 times every week for 6 weeks.
  Interventions: Dietary Supplement: Very low calorie diet (VLCD); Other: Resistance exercise training (RET)
- VLCD+HIIT (Active Comparator): VLCD+HIIT group- participants in this group will receive complete meal replacement for 6 weeks and High intensity interval training 3 times every week for 6 weeks.
  Interventions: Dietary Supplement: Very low calorie diet (VLCD); Other: High intensity interval training (HIIT)

INTERVENTIONS:
Dietary Supplement: Very low calorie diet (VLCD) — All participants (including exercise group) will be using full daily meal replacement during the 6-week interventional period. The total meal supplement is 600 kcal/day.
  Other Names: LighterLife meal replacement
Other: High intensity interval training (HIIT) — Participants in this group will be having HIIT session three times per week under close medical supervision. This involves 60 sec high intensity cycling at 95-125% Watt Max, with 90s recovery, repeated 5 times, with 2 minutes warm up and cool down.
  Arms: VLCD+HIIT
Other: Resistance exercise training (RET) — The exercise format will be 2 sets of 12 repetitions at 70% 1-RM for each resistance regime, with 1-2 minutes rest between sets after a prescribed warm-up 3 sessions/week. The resistance regimes are: (3 upper body)chest press, latissimus pull down, seated lever row; (3 lower body) leg extension, leg curl, leg press. Participants will be alternating between upper and lower body exercise during each training session.
  Other Names: Weight training
  Arms: VLCD+RET

SUMMARY:
The aims of this project are: to investigate the impact of VLCD on control of muscle protein synthesis, muscle structure and function, cardiac function (ejection fraction), vascular function (blood flow and capillary function), overall physiology status (cardiopulmonary function) and metabolic status (insulin sensitivity) in overweight and obese middle-aged male with or without exercises.

There are 3 groups for the study, to which each participant will be randomly assigned into one of either:

1. VLCD only
2. VLCD with resistance exercise training (RET)
3. VLCD with high intensity interval training (HIIT) The total duration of the intervention is six weeks, with exercises taking place three times per week at the research unit under close supervision by trained staff.

DETAILED DESCRIPTION:
Recent interest has emerged on the role of hypoenergetic very low calorie diets (VLCD) in managing overweight and obese people with or without type 2 diabetes. However, VLCD results in 20-30% of mass lost as lean body mass (LBM) besides adipose tissue. Since LBM in the form of skeletal muscle plays an important role for maintaining whole-body metabolic health and represents a vast protein store, better understanding of the mechanisms of VLCD induced weight loss is very important. In a recent systematic review, the investigators observed that information on the subject is scarce. Early studies with VLCD, using poor quality protein supplements showed that VLCD was associated with an increased risk of adverse mortality outcome mainly due to cardiac muscle atrophy. Although current VLCDs are safer, concerns regarding preservation of LBM persist. This is because, in middle-aged (and older) people who are already suffering the early stages of sarcopenia at approximately 0.5-1%/y from the age of ~40y, VLCD may result in additional significant muscle mass loss. Low muscle mass, especially in older individuals is associated with increased mortality, dynapenia (reduced muscle function) and numerous metabolic conditions. Exercises remain the most effective means by which to maintain and increase muscle mass through stimulation of muscle protein synthesis (MPS). Although studies have shown that losses of LBM during a VLCD can be attenuated with the inclusion of resistance exercise training (RET) [5], the mechanism by which VLCD (with and without exercise) effects MPS is poorly defined. The investigators also know now that high intensity interval training (HIIT) improves LBM, cardiac and metabolic function, yet no study has clarified the outcome of HIIT with VLCD on MPS and LBM. The investigators will investigate the different effects of VLCD with RET, VLCD with HIIT, and VLCD alone on MPS and overall metabolic function in overweight middle-aged males.

This project aims to investigate the impact of VLCD on MPS, insulin sensitivity, muscle structure and function (strength), cardiopulmonary fitness in overweight and obese middle-aged adults with or without RET or HIIT. The investigators hypothesised that VLCD will impair MPS and slightly reduce muscle thickness and function, and cardiopulmonary fitness, while exercises will improve MPS and muscle structure and function. All group will show overall improve in insulin sensitivity.

This study will involve 36 overweight (and obese) male (BMI 27-50kg/m2) subjects aged 30-60y. Subjects will be randomised into one of 3 groups (12 each) following baseline investigations and prior to starting interventions: 1) VLCD; 2) VLCD + RET; 3) VLCD + HIIT.

Subjects will be excluded if they have evidence of:

* Participation in a formal exercise regime
* Active cardiovascular disease: uncontrolled hypertension (BP > 180/110), angina, heart failure (class III/IV), arrhythmia, right to left cardiac shunt, recent cardiac event
* Cerebrovascular disease: previous stroke, aneurysm (large vessel or intracranial), epilepsy
* Respiratory disease including: pulmonary hypertension, chronic obstructive pulmonary disease (COPD), severe uncontrolled asthma,
* Diabetes mellitus.
* Active inflammatory bowel or renal disease
* Malignancy
* Clotting dysfunction
* Musculoskeletal or neurological disorders
* Family history of early (<55y) death from cardiovascular disease
* Known sensitivity/ allergy to contrast Sonovue
* Any other ongoing acute or significant chronic medical condition that is not mentioned above.
* Weight >120kg -weight limit for dual energy x-ray absorptiometry (DXA) scan All subjects will undergo a full medical screening before being enrolled into the study. This screening will involve measures of height and weight, medical history and physical examination, blood tests (for fasting FBC's, U&E's, LFT's, TFT's, glucose, HbA1C, lipid profiles and coagulation), and ECG. Abnormal screening results will be discussed with the subject and their General Practitioner (GP) will be informed appropriately.

Subject who meets inclusion criteria will be enrolled and randomised to one of the 3 groups (outlined above) and invited to attend for baseline investigations (before intervention). Subjects will be asked to fast from midnight (except clear water) prior to attending their first day of investigations: DAY(-4). On this day, baseline investigations will include a DXA scan, fasting specimen (blood glucose, saliva, muscle and fat) collection, vascular ultrasound scans (flow mediated dilation (FMD), leg blood flow (LBF)), and an oral glucose tolerance test (OGTT) with 2-Deoxyglucose (2DOG) tracer infusion to assess glucose uptake and insulin sensitivity. The muscle biopsy will be repeated after the 2DOG infusion, followed by leg ultrasound scans to assess muscle structure. A standard lunch will be provided in the afternoon. A cardiac echocardiogram (ECHO) will be performed to assess cardiac function followed by ultrasound scan (USS) of dominant thigh muscles (for pennation angle, thickness, fascicle length) and cardiopulmonary exercise test (CPET) to determine maximal aerobic capacity and set the load for the HIIT training (Watt Max, where applicable). A loading dose of deuterium oxide (D2O) and D3 creatine tracer solutions will then be given. Before leaving, subjects will be supplied with 3-Methylhistidine (3MH) tracer solution to be taken 2 days later DAY(-2), plus daily 'top-ups' of D2O (all tracer amounts based on body weight). Saliva bottles for daily saliva collection (3 hours after daily D2O top up, to be stored in the fridge) and containers for urine collection for D3 creatine assessment (daily urine sample collection for 3 days in containers begin with 24-hour urine collection, then spot urine at 30h, 48h and 72h) for muscle mass assessment will also be provided. After consuming 3MH on DAY(-2), subjects will then attend our unit the next day (DAY(-1)) in the morning, fasted from midnight (except clear water). Hourly blood samples for 6 hours to measure 3MH levels (the first sample to be taken 20-24 hours after 3MH ingestion) and contrast enhanced ultrasound (CEUS) will be done. Following this, baseline muscle strength/ function will be assessed; 1 repetition maximum (1-RM) assessment on 6 (3 upper body, 3 lower body) exercises and maximal voluntary contraction (MVC) of leg extension. After this visit subjects will begin their intervention period (DAY 1) according to their group. All groups will have a 6-week intervention period of nutritional intervention in the form of LighterLife VLCD meal replacement diets: 4 meals/day providing 600kcal/d with 100% recommended daily allowance (RDA) vitamins and minerals. For RET group, the exercise format will be 2 sets of 12 repetitions at 70% 1-RM for each muscle group with 1-2 minutes rest between sets after a prescribed warm-up 3 sessions/week. The exercises will involve upper and lower body exercises and will be progressive in nature with muscle strength assessed every ~14 days to ensure that the intensity of training remains constant throughout. In the HIIT group, it will be 3 sessions/week, involving 60s high intensity cycling at 95-125% Watt Max, with 90s recovery, for 5 cycles, with 2 minutes warm up and cool down. All subjects will have blood samples (including 3MH tracer) and muscle/ fat biopsies every 3 weeks. DXA scan, ultrasound measurements (vascular and muscle), D3 creatine assessment, 2DOG infusion, OGTT (as explained above), CPET, MVC, muscle strength assessment will be performed before and after the 6-week intervention period. Subjects will be collecting saliva daily into saliva bottles. The collections will be kept in fridge and will be sent to our unit 3 times/week for exercise group (during exercise sessions), and once a week for VLCD only group. Diet diary and physical activity (Actiheart Monitor) also will be monitored (for 4-5 days) before and during interventions, which should include weekend measurement.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age 30 to 60-year old
* BMI 27 to 50

Exclusion Criteria:

* Participation in a formal exercise regime more than 2 hours, twice per week
* Active cardiovascular disease: uncontrolled hypertension (BP > 180/110), angina, heart failure (class III/IV), arrhythmia, right to left cardiac shunt, recent cardiac event
* Cerebrovascular disease: previous stroke, aneurysm (large vessel or intracranial), epilepsy
* Respiratory disease including: pulmonary hypertension, COPD, severe uncontrolled asthma,
* Diabetes mellitus.
* Active inflammatory bowel or renal disease
* Malignancy
* Clotting dysfunction
* Musculoskeletal or neurological disorders
* Family history of early (<55y) death from cardiovascular disease
* Known sensitivity/ allergy to contrast Sonovue
* Any other ongoing acute or SIGNIFICANT chronic medical condition that is not mentioned above.
* Weight >120kg (weight limit for DXA scan)

Ages: 30 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male gender
Enrollment: 36 (Estimated)
Dates: Start 2017-01-09 (Actual); Primary Completion 2019-05-31 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Assessment muscle protein synthesis (MPS) using fractional synthesis rate (FSR) | Baseline, 3 week (midpoint) and post (6-week) intervention
  FSR is calculated from the new alanine incorporation into muscle tissue (from muscle biopsy) in comparison to total D2O body water enrichment over a period of time. The total body D2O enrichment will be assessed from saliva collection, pre and post D2O consumption (few samples per week). As the investigators are planning for daily D2O top-up, the enrichment level hopefully would be stable within a certain level.

SECONDARY OUTCOMES:
Muscle protein breakdown (MPB) | Baseline, 3 week (midpoint) and post (6-week) intervention
  Muscle protein breakdown (MPB) will be assessed using 3-Methylhistidine (3MH) blood and urine sample.
Lipids profile | Baseline, 3 week (midpoint) and post (6-week) intervention
  Blood will be taken to measure changes in lipid profile
Total body skeletal muscle mass | Baseline and post 6-week intervention
  Total body skeletal muscle mass will be assessed using D3-creatine by measuring enrichment of urine D3-creatinine
Total lean body mass | Baseline and post 6-week intervention
  Analysis of changes in total lean body mass (in comparison to fat mass) using DXA scan
Muscle structure | Baseline and post 6-week intervention
  Using USS, structure of vastus lateralis muscle of the dominant leg will be assessed
Muscle strength using 1-RM conversion | Baseline and post 6-week intervention
  3 upper and 3 lower limbs movement will be assessed for strength (Chest press, Latissimus-pull down, Seated lever row, Leg extension, Leg curl, Leg press) using 1-RM conversion following weight assessment.
Maximum voluntary contraction (MVC) of dominant knee extension | Baseline and post 6-week intervention
  Maximal voluntary contraction (MVC) of dominant knee extension will be assess using our standard dynamometer.
Insulin resistance | Baseline and post 6-week intervention
  Insulin resistance will be assessed using homeostasis model assessment (HOMA) formula
Insulin sensitivity | Baseline and post 6-week intervention
  Insulin sensitivity will be assessed via 2 hour OGTT involving blood sampling every 15 minutes for glucose and insulin level measurement.
Assessment of vascular endothelial function using FMD | Baseline and post 6-week intervention
  Flow-mediated dilation (FMD) will be used to assess endothelial function
Blood perfusion to vastus lateralis | Baseline and post 6-week intervention
  Contrast-enhanced ultrasound (CEUS) will be used to assess blood perfusion of the vastus lateralis muscle of dominant leg at rest and following exertion (6 reps of 50% 1-RM knee extension)
Leg blood flow | Baseline and post 6-week intervention
  Leg blood flow (via femoral artery) of dominant leg will be assessed using USS at rest aand in response to acute stimulant (ie 6 repetitions of 50% 1-RM knee extension)
Cardiopulmonary fitness | Baseline and post 6-week intervention
  CPET will be used to assess aerobic threshold.
Cardiac systolic function | Baseline and post 6-week intervention
  ECHO will be used to assess systolic ejection fraction.

CONTACTS AND LOCATIONS:
Overall Officials: Iskandar Idris, Principal Investigator — University of Nottingham
Locations (1):
- MRC-ARUK Centre of Excellence for Musculoskeletal Ageing, School of Medicine, University of Nottingham,, Derby, Derbyshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
No specific plan yet for data sharing.